CLINICAL TRIAL: NCT02434510
Title: Bacterial Contamination of Operative Splash Basins: Can it be Prevented?
Brief Title: Bacterial Contamination of Operative Splash Basins
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jeremy Gililland, M.D., University of Utah
Other Study IDs: 76754
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Infection
Keywords: Infection; Total Knee Arthroplasty; Total Hip Arthroplasty; Splash Basins
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sterile Water bath: Standard of Care group using a sterile water instrument bath
- CHG group: Study group using the 0.05% CHG solution in the instrument bath

SUMMARY:
The primary objective of this study is to compare the efficacy of adding 0.05% chlorhexidine gluconate to the splash basin in reducing bacterial growth from splash basins at the end of a total joint replacement procedure.

Hypothesis: The 0.05% chlorhexidine gluconate solution will reduce the bacterial growth at the end of elective total joint arthroplasty cases.

Null Hypothesis: There will be no difference in bacterial growth from the splash basin at the end of the case despite the addition of an antimicrobial solution.

DETAILED DESCRIPTION:
Total joint arthroplasty of the hip and knee is a procedure growing substantially in number in the United States. Projections approach 2 million combined total hip and total knee arthroplasty procedures by the year 2021[1, 2]. With the incidence of post-arthroplasty infection ranging from 1-2% of primaries and 3-5% of revisions, the number of cases of periprosthetic infection will be significant[1, 3-7]. The associated economic burden is projected to exceed $1.62 billion[2]. With these numbers in mind it is our responsibility in the orthopaedic community to do what we can to reduce the social and economic impact that this devastating complication creates.

While all surgical procedures carry the risk of bacterial contamination, those that implant prosthetic material are particularly high risk for future problems due to the development of biofilms and difficulty eradicating such infections. The most common time of inoculation of the implant is at the time of surgery. Whyte et al.[8] showed that the source of infection was the operating room personnel in 98% of cases while only 2% of the time it was the patient's own skin. The transfer of contaminants occurred via direct transfer through the hands or instruments 70% of the time. Knobben et al.[9] reported transfer of bacteria between biomaterial surfaces at a rate of 17%-71% demonstrating the ability of bacteria to spread to all types of materials in the operative field. The direct contact of these surfaces with the patient or prosthetic implant makes early contamination during surgery a likely cause of periprosthetic infection. Maathuis et al.[10] suggested that at least 30% of patients leave the operating suite with bacterial contamination.

The splash basin has been used for many years in the operating room as a place to wash instruments and clean them of debris for potential re-use during the surgical case. This often places multiple instruments within the bath of washings or in direct contact with previously used tools. Several studies have shown evidence of bacterial contamination of these basins[11-14]. Rates of 2.17% to 74% of contamination of the splash basin have been reported. In a study by Anto et al.[11] an average of 45.7 instruments were placed in the splash basin per case. The opportunity for bacteria to be transferred to the surgical wound upon re-use of an instrument from the basin is therefore concerning.

Given that the splash basin is a potential source of surgical wound contamination we have sought to eliminate the bacterial colonization of this source through the addition of an antimicrobial solution to the normal sterile water bath. To compare potential interventions, a prospective study comparing a 0.05% chlorhexidine gluconate (CHG) antimicrobial solution to the current standard of sterile water as a control is proposed. This concentration of CHG followed by a saline rinse has been shown to decrease the risk of infection during wound irrigation without increasing the risk of adverse effects[15, 16].

Given our expertise in the area of total joint arthroplasty and experience with treating periprosthetic infections as well as familiarity with various antimicrobial solutions we feel well qualified to perform this study. The results of this study could improve patient outcomes by potentially eliminating a source of infection in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Splash Basins will be selected from primary total joint arthroplasty cases and then randomized to a solution of either sterile water or sterile water with 0.05% CHG.
* Other than being scheduled for a primary total joint arthroplasty, the participant information will not be reviewed for selection of the splash basin, but will be collected for comparison of patient characteristics and potentially for future reference to compare infection rates in patients associated with this study.

Exclusion Criteria:

* Splash basin used in a revision total joint procedure
* Splash basin used in cases where the patient has a history of known periprosthetic joint infection
* Splash basin used in cases where the patient has a known allergy to chlorhexidine gluconate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for primary total joint arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Bacterial Contamination | up to 1-3 days
  After 1-3+ days, agar plates (cultured with splash basin solution) will be pulled from incubation and examined for growth. Basins with any growth of aerobic organisms will be considered as a positive finding.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Gililland, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States